CLINICAL TRIAL: NCT00652327
Title: A Multicenter, Randomized, Open-labeled, Parallel Group Comparison Study to Evaluate the Efficacy, Safety and Tolerability of Ezetimibe Added to Ongoing Statin Therapy Versus Doubling the Dose of Ongoing Statin in the Treatment of Hypercholesterolemia.
Brief Title: Comparison of Ezetimibe Added to Ongoing Statin Therapy Versus Doubling the Dose of Statin in the Treatment of Hypercholesterolemia (P04355)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04355
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2010-06-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Atorvastatin; Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe + Statin (Experimental)
  Interventions: Drug: Ezetimibe + Statin (simvastatin, atorvastatin, or pravastatin)
- Double Statin (Active Comparator)
  Interventions: Drug: Double Statin (simvastatin, atorvastatin, or pravastatin)

INTERVENTIONS:
Drug: Ezetimibe + Statin (simvastatin, atorvastatin, or pravastatin) — ezetimibe 10 mg plus ongoing statin (simvastatin 20 mg or atorvastatin 10 mg or pravastatin 20 mg) once daily for 8 weeks
  Arms: Ezetimibe + Statin
Drug: Double Statin (simvastatin, atorvastatin, or pravastatin) — simvastatin 40 mg or atorvastatin 20 mg or pravastatin 40 mg once daily for 8 weeks
  Arms: Double Statin

SUMMARY:
This is a randomized, open label, parallel group comparison study. Following a 1-week screening period, patients will be randomized to 1 of 2 treatment groups: ezetimibe added to ongoing statin treatment (ezetimibe plus simvastatin, atorvastatin or pravastatin at doses of 10/20, 10/10 or 10/20 mg), or doubling the dose of ongoing statin (simvastatin 40 mg, atorvastatin 20 mg, or pravastatin 40 mg). Study drug will be administered once daily in the evening for 8 weeks. Patients will be instructed to follow a National Cholesterol Education Program (NCEP) or similar cholesterol-lowering dietary regimen throughout the study.

ELIGIBILITY:
Inclusion Criteria:

80-120 patients will be recruited in this study. All patients must meet the following criteria and follow an NCEP or similar cholesterol-lowering dietary regimen throughout the study:

* Men or women ≧18 and ≦80 years of age (Female patients receiving hormone therapy [including hormone replacement therapy, and estrogen antagonist/agonist, or oral contraceptives] and maintained on a stable dose and regimen for at least 8 weeks prior to visit 1 must be willing to continue the same regimen throughout the study. Females of childbearing potential must be using a medically acceptable method of birth control).
* Willing to follow an NCEP Therapeutic Lifestyle Changes (TLC) or similar cholesterol-lowering diet for the duration of the study.
* Patients with hypercholesterolemia who cannot achieve the optimal therapeutic goal with previous statin treatment (simvastatin 20 mg, atorvastatin 10 mg or pravastatin 20 mg alone for at least 12 weeks) will be enrolled into study. The treatment goal in primary prevention is LDL-C <160 mg/dL or LDL-C <130 mg/dL patient with ≧ 2 risk factors (risk factors: hypertension, male ≧ 45 years old, family of premature coronary artery disease [CAD], female ≧ 55 years old or menopause without hormone replace therapy, smoking); LDL-C ≤ 100 mg/dL in CAD patients (documented by coronary angiogram, positive treadmill test or thallium scan), or diabetes mellitus (DM) patients (Ante Cibum [AC][fasting plasma glucose] >126 mg/dL, Post Cibum [PC] [oral glucose tolerance test] > 200 mg/dL, World Health Organization criteria), ischemic stroke (neurological dysfunction with documented diagnosis with computed tomography [CT] or magnetic resonance imaging [MRI]), peripheral artery disease.
* Triglyceride (TG) concentrations ≦ 400 mg/dL.
* Liver transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) ≦ 2 x upper limit of normal (ULN) with no active liver disease and creatine kinase (CK) ≦ 2 x ULN at screen visit.

Exclusion Criteria:

The following conditions preclude patients from entry into this study:

* Women who are pregnant or lactating.
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy
* Patients who have been treated with any other investigational drug within 3 months of visit 1.
* Patients previously randomized to a study with ezetimibe.
* Active liver disease or Impaired liver function tests (ALT, AST > 2xULN).
* Impaired renal function ( serum creatinine ≧1.5 mg/dL) or nephrotic syndrome at visit 1
* Unstable angina
* Acute myocardial infarction, coronary bypass surgery within the previous six months of visit 1.
* Uncontrolled cardiac arrhythmias
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure > 160 mmHg or diastolic > 100 mmHg at visit 1.
* Poorly controlled diabetes mellitus patient (Patients who are under insulin injection and HbA1c>10.0%). If the patient is treated with medication for diabetes, the medication will be unchanged during the study period.
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoprotein, e.g. hypothyroidism (thyroid-stimulating hormone [TSH] > 5.5 uIU/mL). However, patients who are on a stable therapy of thyroid replacement therapy for at least 6 weeks are eligible for enrollment.
* Patients hypersensitive to HMG-CoA reductase inhibitors or ezetimibe.
* Patient who is unable to give informed consent (the patient with a legal representative to sign the informed consent is eligible to participate the study).
* Any condition or situation which, in the opinion of the investigator, might pose a risk to the patient or confound the results of the study.
* Prohibited concomitant therapies.

  * Medications that are potent inhibitors of CYP3A4, including cyclosporine, systemic itraconazole or ketoconazole, erythromycin or clarithromycin, nefazodone, verapamil and human immunodeficiency virus (HIV) protease inhibitors.
  * Lipid-lowering agents including fish oils, Cholestin, bile-acid sequestrants, and niacin (<200 mg/day) taken within 6 weeks and fibrates taken within 8 weeks prior to enrollment.
  * Oral corticosteroids unless used as replacement therapy for pituitary/adrenal disease and treated with a stable regimen for at least 6 weeks prior to enrollment.
  * Treatment with psylium, other fiber-based laxatives, and/or over-the-counter (OTC) therapies known to affect serum lipid levels, phytosterol margarines, unless treated with a stable regimen for at least 6 weeks prior to enrollment, and patient agrees to remain on constant regimen for the duration of the study.
* Patient is consuming > 250 ml of grapefruit juice per day.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

REFERENCES:
- [Derived] Yu CC, Lai WT, Shih KC, Lin TH, Lu CH, Lai HJ, Hanson ME, Hwang JJ. Efficacy, safety and tolerability of ongoing statin plus ezetimibe versus doubling the ongoing statin dose in hypercholesterolemic Taiwanese patients: an open-label, randomized clinical trial. BMC Res Notes. 2012 May 23;5:251. doi: 10.1186/1756-0500-5-251. PMID 22621316

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 202 potential participants signed informed consent during a screening visit. Of these, 119 did not meet protocol eligibility requirements. The remainder, 83, received randomized treatment assignment.
Groups:
- Ezetimibe + Statin: Once daily 10-mg ezetimibe tablet added to daily ongoing statin treatment (simvastatin 20 mg or atorvastatin 10 mg or pravastatin 20 mg) for 8 weeks
- Double Statin: Double the dose of daily ongoing statin treatment (simvastatin 20 mg or atorvastatin 10 mg or pravastatin 20 mg) for 8 weeks
Period: Overall Study
Arm/Group | Ezetimibe + Statin | Double Statin
Started | 42 (Participants who recieved randomized treatment assignment to ezetimibe and ongoing statin) | 41 (Participants who recieved randomized treatment assignment to double the dose of ongoing statin)
Completed | 42 | 36
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe + Statin | Double Statin | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 83 years | 42 | 41 | 83
  >=83 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 23 | 23 | 46
Region of Enrollment [Number; unit: Participants]
  Taiwan, Province Of China | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline at Study Endpoint, After 8 Weeks of Treatment
Time Frame: Assessed at the end of 8 weeks of treatment (from baseline to endpoint)
Population: The population analyzed (intent-to-treat [ITT]) included all participants who had a post-randomization LDL-C laboratory evaluation. As such, 20 of the 83 participants who received treatment assignment were excluded from the ITT. The 5 participants who discontinued were included in the ITT as each had a post-randomization LDL-C lab evaluation.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ezetimibe + Statin | Double Statin
Number analyzed (Participants) | 29 | 34
Percentage change | -26.56 (19.78) | -9.7 (21.07)
Statistical Analysis 1: Comparison: Ezetimibe + Statin vs Double Statin; Test type: Superiority or Other; p = .0026, Wilcoxon rank sum test

ADVERSE EVENTS:
Arm/Group | Ezetimibe + Statin | Double Statin
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe + Statin (N=42) | Double Statin (N=41)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe + Statin (N=42) | Double Statin (N=41)
vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less